CLINICAL TRIAL: NCT01032590
Title: Internet Weight Loss Intervention for Individuals Diagnosed With Colorectal Cancer
Brief Title: Internet-Based Weight-Loss Program for Colorectal Cancer Survivors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial was only opened at RCINJ for analysis of data, no patient enrollment took place here.
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 130902; P30CA072720 (NIH); CDR0000660594 (Other: NIH)
Record Dates: First submitted 2009-12-13; First posted 2009-12-15 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Cancer Survivor; Colorectal Cancer; Weight Changes
Keywords: weight changes; cancer survivor; stage I colon cancer; stage II colon cancer; stage III colon cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Body Weight Changes; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Arm I (12-week Internet-based weight-loss intervention): After a baseline evaluation, subjects will start a 12 week Internet-based weight-loss intervention.
  Interventions: Behavioral: Internet weight loss intervention
- Arm II (Active Comparator): Arm II (wait-list control): Patients are instructed to continue their usual dietary and physical activity routines during a 12-week wait period. After the waiting period, patients receive the Internet-based weight-loss intervention for 12 weeks as in arm I.
  Interventions: Behavioral: Internet weight loss intervention

INTERVENTIONS:
Behavioral: Internet weight loss intervention — Participants will be advised to login to the website twice a week during the intervention period. They will be prompted to report their weight, to review and update their reasons for weight loss, to indicate their success with implementing each of their weight loss strategies, to rate the perceived effectiveness of each weight loss strategy,and to revise or create new strategies, as needed.

SUMMARY:
RATIONALE: A personalized Internet-based weight-loss program may help improve the quality of life for colorectal cancer survivors.

PURPOSE: This randomized phase I trial is studying how well an Internet-based program works in helping colorectal cancer survivors lose weight.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the feasibility of implementing an Internet-based weight-loss intervention for colorectal cancer (CRC) survivors.
* To obtain preliminary outcome data on the impact of an Internet-based intervention on weight loss, waist circumference, physical activity, diet, weight-control strategies, weight-loss intention, exercise and diet self-efficacy, and perceived weight-loss barriers among CRC survivors.
* To obtain preliminary data on potential moderators (sociodemographics, disease and treatment characteristics, prior Internet experience, depressive symptoms, dieting and weight-loss experiences, weight-loss expectations, and physical activity and dietary outcome expectancies) of weight loss among CRC survivors using an Internet-based weight-loss intervention.

OUTLINE: Patients are stratified according to time since completion of cancer treatment (1 to 2 years vs 3 to 4 years vs 5 to 6 years vs 7 to 10 years). Patients are randomized to 1 of 2 intervention arms.

* Arm I (12-week Internet-based weight-loss intervention): Patients attend an in-person 60-minute session with a health educator. The health educator will review the patient's weight history, current eating habits, prior and current level of physical activity, reasons for wanting to lose weight, current weight, weight-loss goals, and barriers to weight loss. The health educator will provide basic weight-loss advice for the patient, according to established guidelines, and advice on diet modification to reduce caloric intake. The health educator will also recommend gradual increases in physical activity and help patients set a realistic target weight to achieve at the end of the 12-week intervention period.

The health educator will introduce the intervention website to the patient and assist the patient in setting up a confidential, unique login username and password that will provide secure access to the study website. Patients are asked to provide an email address. After logging onto the website and viewing an introductory page, patients are prompted to specify their target weight for the end of the 12-week intervention and to provide a list of reasons for wanting to lose weight. Next, the website prompts patients to list specific strategies that they plan to use to achieve their desired weight loss. The health educator will guide the patient in entering an initial set of strategies and will provide the patient a list of examples of weight-loss strategies and encourage the patient to generate his/her own specific, personalized strategies. Patients will also be able to select and adapt strategies from the example list that they feel are appropriate for them. The health educator will ensure that the patient is comfortable using the website and will give the patient a one-page written summary of how to use the website and a phone number and an e-mail address that they can use to receive technical help with the website. Additionally, patients are advised to login to the website twice a week during the 12-week intervention period and are prompted to report their weight, to review and update their reasons for weight loss, to indicate their success with implementing each of their weight-loss strategies, to rate the perceived effectiveness of each weight-loss strategy, and to revise or create new strategies as needed. Patients will also receive automated e-mails that prompt them to visit the website and that provide them with weight-loss tips and motivational messages. The website also provides additional resources, including a list of credible external websites with useful weight loss information and healthy recipes, a summary of weight-loss tips, tips for creating appropriate weight-loss strategies, and examples of weight-loss strategies.

* Arm II (wait-list control): Patients are instructed to continue their usual dietary and physical activity routines during a 12-week wait period. After the waiting period, patients receive the Internet-based weight-loss intervention for 12 weeks as in arm I.

Patients in both arms complete surveys at baseline and at 12 weeks to assess sociodemographics, disease and treatment characteristics, prior Internet experience, depressive symptoms, weight, dieting and weight-loss experiences, weight-loss expectations, and physical activity and dietary outcome expectancies. Patients in arm II also complete an additional follow-up survey at 24 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of colorectal cancer (CRC)

  * Stage I-III disease
* Completed treatment for CRC 1-10 years ago
* No current evidence of cancer

PATIENT CHARACTERISTICS:

* Not nursing
* Not pregnant within the past 6 months and not planning to become pregnant
* Speaks English
* Has access to the Internet at home or work
* Lives within 50 miles of Fox Chase Cancer Center (FCCC)
* Body mass index 25 to 35 kg/m^2
* No weight loss of ≥ 15 lbs within the past 6 months
* No history of eating disorder
* None of the following medical conditions:

  * Myocardial infarction or stroke within the past 6 months
  * Type I diabetes
  * Uncontrolled hypertension
  * Unstable angina
  * Congestive heart failure

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent weight-loss medications (intervention phase)

Ages: 21 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2017-03-02 (Actual); Study Completion 2017-03-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of implementing an Internet-based weight-loss intervention for colorectal cancer survivors | 5 years
Impact of an Internet-based intervention on weight loss | 5 years

SECONDARY OUTCOMES:
Impact of an Internet-based intervention on waist circumference, physical activity, diet, weight-control strategies, weight-loss intention, exercise and diet self-efficacy, and perceived weight-loss barriers | 5 years
Potential moderators of weight loss | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Coups, PhD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (2):
- United States (2):
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania